CLINICAL TRIAL: NCT00001108
Title: Multi-Drug Antiretroviral Therapy for Heavily Pretreated Pediatric AIDS Patients: A Phase I Proof of Concept Trial
Brief Title: A Study of the Safety and Effectiveness of Treating Advanced AIDS Patients Between Ages 4 and 22 With 7 Drugs, Some at Higher Than Usual Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: P1007; 11643 (Registry Identifier: DAIDS ES); ACTG P1007; PACTG P1007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Salvage Therapy; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Saquinavir; Nevirapine; Lamivudine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Saquinavir
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if 7 drugs, some of them given at higher doses than normal, are safe and tolerated by young patients with AIDS who have failed to respond to other treatments. The study will also see what effect taking several anti-HIV drugs together at high doses has on the body's ability to fight HIV infection. The 7 drugs that will be given in this study are stavudine (d4T), didanosine (ddI), lamivudine (3TC), nelfinavir (NFV), ritonavir (RTV), saquinavir (SQV), and nevirapine (NVP).

(This study has been changed from an 8-drug regimen to a 7-drug regimen. Patients no longer receive the drug hydroxyurea [HU].) Doctors are seeing many HIV-positive children who did not get good long-term results from the current anti-HIV drugs. Some doctors believe anti-HIV drugs fail because drug levels in the body are too low. In this study, doctors will give patients 7 drugs, some at higher doses than normal. Since it is very important that patients on the study take all of these drugs, doctors will make it as easy as possible. Doctors want to try this because children with advanced AIDS have few treatment choices.

DETAILED DESCRIPTION:
Clinicians are increasingly confronted with HIV-positive children who have failed all available antiretroviral therapies and have few viable treatment options. Virologic failure in these patients may be a result of antiretroviral resistance, likely a result of poor adherence to the treatment regimen or inadequate dosing. This study is designed to achieve adherence through observation of drug administration for the first 8 weeks of the study and to further overcome resistance by intensive, high-dose, multi-drug therapy. Treatment with more than 4 drugs has not been studied formally in children, but pediatricians caring for children with AIDS have used such strategies off study with success. Dose intensification may also aid in overcoming resistance; therefore, in this trial, d4T, 3TC, and NFV are administered at up to twice their standard doses. Given the limited therapeutic options available to HIV-positive children with poor prognoses, high-dose, multi-drug therapy merits study. [AS PER AMENDMENT 01/07/00: Pancreatitis, which may be fatal in some cases, has occurred during therapy with ddI. The risk of pancreatitis may be increased when ddI is used in combination with HU. ACTG A5025, a study that had a d4T/ddI/HU arm, was terminated because of significant toxicity concerns related to the HU-containing arm. Patients enrolled in ACTG P1007 may be at increased risk of developing pancreatitis given their advanced disease state and the use of multiple drugs including HU. The study had been amended to address these concerns.] [AS PER AMENDMENT 12/19/01: HU has been removed from the drug regimen.]

Patient enrollment is staged to allow study physicians to aggressively monitor patients for signs of toxicity. Initially, patients are admitted to a hospital or clinical research center for 2 weeks, where they initiate an [AS PER AMENDMENT 12/19/01: "8-drug regimen" is replaced by "7-drug regimen"] and undergo frequent physical exams and blood tests to assess [AS PER AMENDMENT 12/19/01: glucose levels], pharmacokinetics, virologic response, and toxicity. If investigators identify important drug interactions requiring modification of the combination regimen, or if there are early regimen-terminating toxicities, the trial will be halted to address these concerns. After 2 weeks, the patient is discharged to return home. Study personnel visit the patient's house twice a day for 6 more weeks to observe drug administration, and the patient continues to receive regular physical exams and blood tests. At the end of Week 24, all patients with plasma RNA levels of 10,000 copies/ml or less are offered the opportunity to continue their regimen to Week 48. Patients with plasma RNA levels above 10,000 copies/ml at Week 24 and patients who experience virologic rebound at or after Week 24 are taken off study unless the patient's family and the investigator feel it is in the best interest of the child to remain on study. [AS PER AMENDMENT 12/19/01: The 2-week hospital or GCRC stay is no longer required. A 2-day stay in a hospital or GCRC for the purpose of drug regimen training is recommended, but not mandatory. Study personnel visit the patient once a day for 6 weeks at an agreed upon location or by phone contact.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this trial if they:

* Are HIV-positive.
* Have HIV levels of 10,000 copies/ml or more.
* Are between ages 4 and 22.
* Have motivation and ability to conform to the complex treatment regimen.
* Agree to practice abstinence or use 2 effective methods of birth control during the study and until 3 months after stopping the study drugs, if sexually active.
* Have written informed consent from a parent or legal guardian if under age 18.
* Have used at least 3 different nucleoside reverse transcriptase inhibitors (NRTIs) for at least 3 months each or have shown resistance to at least 3 different NRTIs.
* Have used at least 1 nonnucleoside reverse transcriptase inhibitor (NNRTI) for at least 3 months each or have shown resistance.
* Have used at least 2 different courses of a protease inhibitor (PI)-containing regimen, each of which was at least 6 months, or have evidence of mutations to at least 2 different PIs.
* This study has been changed. The inclusion criteria reflects a change in the prior anti-HIV therapy required, age requirement, and the required CD4 and HIV levels.

Exclusion Criteria

Patients will not be eligible for this trial if they:

* Are allergic to even 1 study drug or have ever had to stop 1 of these drugs because of a bad reaction to it.
* Have a history of diabetes, hepatitis C, hepatitis B, or certain diseases of the nervous system, heart, or pancreas.
* Have had a serious infection within 14 days of starting the study.
* Need certain drugs that interact with the study drugs. (See Technical Summary for more details.)
* Are pregnant or breast-feeding.
* Have had hepatitis within 30 days of study entry.

Ages: 4 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6
Dates: Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Aldrovandi, Study Chair; Paul Palumbo, Study Chair
Locations (19):
- United States (19):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Univ of Miami (Pediatric), Miami, Florida
  - Sacred Heart Children's Hosp / CMS of Florida, Pensacola, Florida
  - Cook County Hosp, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - North Shore Univ Hosp, Great Neck, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Med College of Virginia, Richmond, Virginia